CLINICAL TRIAL: NCT00991068
Title: An Open-Label Pilot Study Evaluating Synera® in the Treatment of Patients With Carpal Tunnel Syndrome
Brief Title: Open-Label Study Evaluating Synera® in the Treatment of Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-201
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Pain; Mild to moderate Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain | interventions — Lidocaine; Tetracaine; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Synera (Experimental): Synera topical patch
  Interventions: Drug: Synera (lidocaine 70 mg and tetracaine 70 mg) topical patch

INTERVENTIONS:
Drug: Synera (lidocaine 70 mg and tetracaine 70 mg) topical patch — Patients will apply a single Synera patch to the target wrist for 2 hours twice a day (ie, morning and evening applications) for 14 days.

SUMMARY:
The purpose of the study is to explore the potential usefulness of Synera for the treatment of pain associated with mild to moderate carpal tunnel syndrome.

DETAILED DESCRIPTION:
ZARS Pharma, Inc. has developed Synera® (lidocaine 70 mg and tetracaine 70 mg topical patch), a drug delivery patch that utilizes controlled heat to enhance the delivery of a local anesthetic formulation consisting of a eutectic mixture of lidocaine and tetracaine. Synera was approved by the Food and Drug Administration (FDA) on June 23, 2005 and is indicated for use on intact skin to provide local dermal analgesia for superficial venous access and superficial dermatological procedures such as excision, electrodesiccation, and shave biopsy of skin lesions.

The purpose of this single center, 2-week open-label pilot study is to explore the potential usefulness of Synera for the treatment of pain associated with mild to moderate CTS.

ELIGIBILITY:
Inclusion Criteria:

* Pain associated with mild to moderate carpal tunnel syndrome in a single wrist
* Have recent (within 3 months) electrodiagnostic evidence of carpal tunnel syndrome (CTS)

Exclusion Criteria:

* Have bilateral carpal tunnel syndrome
* Have another peripheral neuropathy in the affected limb
* Have had an injection into the carpal tunnel within 8 weeks
* Have had surgical release of the target wrist within previous 6 months
* Have electrodiagnostic evidence of severe CTS

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Screening/Day 1, Day 8, and Day 15 or early withdrawal

SECONDARY OUTCOMES:
Pain interference with activities (general, normal work, sleep) | Screening/Day 1, Day 8, and Day 15 or early withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Nalamachu, MD, Principal Investigator — International Clinical Research Institute
Locations (1):
- International Clinical Research Institute, Overland Park, Kansas, United States